CLINICAL TRIAL: NCT05350969
Title: Phase 2, Multicenter, Randomized, Parallel, 3-arm, Placebo-controlled Study to Assess Efficacy and Safety of CDR132L in Patients With Reduced Left Ventricular Ejection Fraction (≤ 45%) After Myocardial Infarction
Brief Title: Study to Assess Efficacy and Safety of CDR132L in Patients With Reduced Left Ventricular Ejection Fraction After Myocardial Infarction
Acronym: HF-REVERT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cardior Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDR132L-P2-01; 2023-507569-24-00 (EU CTIS Number); 2021-006040-27 (EudraCT Number)
Record Dates: First submitted 2022-04-20; First posted 2022-04-28 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Myocardial Infarction, Acute; Heart Failure, Left Sided
MeSH Terms: conditions — Myocardial Infarction; Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Pharmacy staff is unblinded. They will hand-over prepared investigational medicinal product (IMP) in light-protected syringe.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CDR132L 5 mg (Experimental): CDR132L 5 mg/kg body weight intravenous in single dose on Day 1, Day 29 and Day 57
  Interventions: Drug: CDR132L
- CDR132L 10 mg (Experimental): CDR132L 10 mg/kg body weight intravenous in single dose on Day 1, Day 29 and Day 57
  Interventions: Drug: CDR132L
- Placebo (Placebo Comparator): Placebo intravenous in single dose on Day 1, Day 29 and Day 57
  Interventions: Drug: Placebo to CDR132L

INTERVENTIONS:
Drug: CDR132L — CDR132L is a synthetic antisense oligonucleotide (ASO) and a selective inhibitor of microRNA-132-3p (miR-132). miR-132 in cardiomyocytes is a central switch affecting the expression of genes that are crucially involved in maladaptive cardiac remodeling, transformation, and pathological cardiac growth (hypertrophy), contributing to adverse cardiac remodeling and heart failure (HF).1-5 Aberrant expression of miR-132 in cardiac cells is causally associated with cardiac remodeling and HF progression.
  Arms: CDR132L 10 mg; CDR132L 5 mg
Drug: Placebo to CDR132L — Placebo to CDR132L
  Arms: Placebo

SUMMARY:
This is a Phase 2, multicenter, randomized, parallel, 3-arm, placebo-controlled study to assess efficacy and safety of CDR132L in patients with reduced Left Ventricular Ejection Fraction (LVEF) (≤ 45%) after myocardial infarction (MI). This study consists of a screening period (to occur at least 3 days after MI diagnosis), a 6-month double-blind period, and a 6-month extension period with the End of Study (EOS) Visit at Day 360/Month 12.

Two dosages of CDR132L will be tested against placebo on their effects on patients, who just had a heart attack in addition to standard care. The aim of the study is to show that CDR132L is safe and effective to improve heart failure in such patients.

ELIGIBILITY:
Main Inclusion Criteria:

1. Male or female patients, aged ≥ 30 to ≤ 80 years at the date of signing informed consent which is defined as the beginning of the Screening Period.
2. Spontaneous acute mycardial infarction (AMI) (type I) based on the universal MI definition with randomization to occur no later than 14 days after index event diagnosis.
3. Patient with a LVEF ≤ 45% as measured by ECHO after MI diagnosis (STEMI or NSTEMI).
4. Patient with previous MI events in history can be included.
5. Patient with body weight of ≤ 120 kg.
6. N-terminal pro B-type natriuretic peptide level ≥ 125 pg/ml and < 8000 pg/ml at screening.
7. Patient with STEMI/NSTEMI who underwent percutaneous coronary intervention for this event.

Exclusion Criteria:

1. A woman of childbearing potential (WOCBP).
2. Patient with HF of non-ischemic origin; e.g., myocarditis, alcoholic cardiomyopathy.
3. Patient with New York Heart Association (NYHA) class IV at screening or randomization.
4. Patient has any planned cardiac intervention (angiogram without angioplasty is acceptable) or any other planned surgery after the Screening Period.
5. Patient has severe valvular heart disease.
6. Patient has systolic BP < 90 mmHg or > 180 mmHg, diastolic BP < 50 mmHg or > 110 mmHg, and/or heart rate < 50 or > 100 beats/minute at screening or randomization.
7. Patient with an estimated glomerular filtration rate < 30 mL/min/1.73 m2 or on dialysis.
8. Patient with hepatic insufficiency classified as Child-Pugh B or C.
9. Patient has medical history of disease(s) affecting the blood-brain-barrier, e.g., stroke within 6 months or multiple sclerosis.
10. Patient has medical history of bleeding disorders or has thrombocytopenia (platelets < 100,000/μL).
11. Patient has poorly controlled diabetes as determined by the Investigator.
12. Patient has a history or presence of any of the following cardiac conditions: known structural cardiac abnormalities beyond HF, family history of long QT syndrome, cardiac syncope, or recurrent, idiopathic syncope.
13. Any clinically significant abnormalities, at the discretion of the Investigator, in rhythm, conduction, or morphology of resting ECG that pose an additional safety risk to patients.
14. Patient with active "severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2)" infection confirmed as per the local testing guidelines at screening.
15. Patient is not to be enrolled into the study if they received any prohibited therapy within 3 months of screening.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2025-03-17 (Actual)

PRIMARY OUTCOMES:
Echocardiography (ECHO) | 6 months
  Percent change from baseline (screening to occur at least 3 days after MI diagnosis as measured by ECHO [central laboratory]) in Left Ventricular End-Systolic Volume (LVESVI) at Month 6.

CONTACTS AND LOCATIONS:
Overall Officials: Johann Bauersachs, Prof. Dr., Principal Investigator — Hannover Medical School
Locations (49):
- Czechia (2):
  - Institut klinicke a experimentalni mediciny, Prague
  - Všeobecná fakultní nemocnice v Praze, Prague
- Germany (8):
  - St. Marien-Krankenhaus Ahaus, Ahaus
  - Herzzentrum Dresden Universitätsklinik, Dresden
  - Helios Klinikum Erfurt, Erfurt
  - Universitätsmedizin Göttingen, Göttingen
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Klinikum Ludwigshafen, Ludwigshafen
  - Universitätsklinikum Würzburg, Würzburg
- Greece (3):
  - "Alexandra" General Hospital of Athens, Athens
  - "Attikon" General University Hospital, Athens
  - General University Hospital of Patras "Panagia i Voitheia", Pátrai
- Semmelweis University, Budapest, Hungary
- Netherlands (10):
  - Jeroen Bosch Ziekenhuis (JBZ) (Hieronymus Bosch Hospital) - locatie Den Bosch, 's-Hertogenbosch
  - Deventer Ziekenhuis, Deventer
  - Slingeland Ziekenhuis, Doetinchem
  - Gelderse Vallei Ziekenhuis, Ede
  - Medisch Centrum Leeuwarden, Leeuwarden
  - St. Jansdal Ziekenhuis, Lelystad
  - Erasmus University Medical Center, Rotterdam
  - Ikazia Ziekenhuis, Rotterdam
  - D & A Research B.V., Sneek
  - Gelre Ziekenhuizen, Zutphen
- Poland (12):
  - Polsko Amerykanskie Kliniki Serca, Kędzierzyn-Koźle
  - Specjalistyczna Poradnia Kardiologiczna i Nadcisnienia Tetniczego, Kielce
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II, Krakow
  - Gabinet Internistyczno-Kardiologiczny Jacek Nowak, Libiąż
  - NZOZ SALUS JZ Peruga, Lodz
  - One wojskowy Szpital Kliniczny w Lublinie, Lublin
  - Medicome Sp. z o.o., Oświęcim
  - Wojewódzki Szpital im. Sw. Ojca Pio w Przemyslu, Przemyśl
  - NZOZ Pro-Cordis Sopockie Centrum Bad. Kardiolog, Sopot
  - Wojewodzki Szpital Zespolony, Torun
  - Spec.Szpital im.dr Sokolowskiego, Wałbrzych
  - Investigational Site, Wroclaw
- Spain (9):
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital de la Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario San Cecilio, Granada
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario de Sabadell, Sabadell
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Complejo Hospitalario Universitario de Vigo, Vigo
- United Kingdom (4):
  - Queen Elizabeth University Hospital, Glasgow
  - Wycombe Hospital, High Wycombe
  - Richmond Pharmacology Limited, London
  - South Tees Hospital NHS Foundation Trust, Middlesbrough

IPD SHARING:
Plan to Share IPD: No